CLINICAL TRIAL: NCT05093530
Title: A Two-part, Randomized, Double-blind, Placebo Controlled, Ascending Dose Study to Assess the Safety and Tolerability of Single and Multiple Doses of Neumifil (a Novel Drug Candidate With Potential for Treatment of COVID-19)
Brief Title: Safety and Tolerability of Single and Multiple Doses of Neumifil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pneumagen Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PNG-NMF-101
Record Dates: First submitted 2021-09-29; First posted 2021-10-26 (Actual); Results first posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Viral Respiratory Tract Infection

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neumifil (Experimental): Neumifil will be administered intranasally using an Aptar delivery system. Each dose will consist of 0.5ml to each nostril, with adjusted concentrations of solution to enable dose ranging. Participants in Part A will receive a single dose of Neumifil and participants in Part B will receive once daily doses of Neumifil for 7 days according to the randomization.
  Ascending single doses for Part A are anticipated to be 0.028mg (group A1), 0.085mg (group A2), 0.28mg (group A3), 0.885mg (group A4) and 2.8mg (group A5). Two further groups of up to 9 subjects may be investigated. The planned dose levels may change following review of the safety and tolerability of previous doses. The maximum dose will not exceed 2.8mg.
  The starting dose level (dose and dose regimen) in Part B will be determined following review of the safety and tolerability of at least 3 dose levels in part A and subsequent dose levels will be determined following review of the safety and tolerability of previous doses.
  Interventions: Drug: Neumifil
- Placebo (Placebo Comparator): Placebo will be administered intranasally using an Aptar deliver system. Each dose will consist of 0.5ml to each nostril. Participants in Part A will receive a single dose of placebo according to the randomization and participants in Part B will receive once daily doses of placebo for 7 days according to the randomization schedule.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Neumifil — Neumifil contains the active ingredient HEX17, a multivalent, glycan-targeting carbohydrate binding module (CBM). HEX17 CBM is suspended in an aqueous buffer solution containing 20 mM sodium phosphate, 50 mM NaCl (at pH 6.3), 5 % (v/v) glycerol and 0.5 % (v/v) polysorbate 80.
  Other Names: HEX17
  Arms: Neumifil
Drug: Placebo — Aqueous buffer solution containing 20 mM sodium phosphate, 50 mM NaCl (at pH 6.3), 5 % (v/v) glycerol and 0.5 % (v/v) polysorbate 80.
  Arms: Placebo

SUMMARY:
This is a Phase 1, single-centre, randomised, placebo-controlled first in human study in healthy subjects. The study will assess the safety and tolerability of single-ascending (Part A) and multiple-ascending (Part B) doses of Neumifil, administered intranasally.

DETAILED DESCRIPTION:
Part A will include up to 36 healthy subjects in up to 5 groups. 6 subjects will be enrolled in Groups A1-A3 and 9 subjects will be enrolled in Groups A4 and A5. All subjects will receive a single intranasal dose of Neumifil or placebo. In Groups A1-A3, 4 subjects will receive Neumifil and 2 will receive matching placebo. In Groups A4 and A5, 6 subjects will receive Neumifil and 3 will receive matching placebo. The planned dose levels are: 0.028 mg (Group A1), 0.085 mg (Group A2), 0.28 mg (Group A3), 0.885 mg (Group A4), and 2.8 mg (Group A5). Additional dose levels may be assessed in up to 2 optional groups of up to 9 subjects each (Groups A6 and A7).

Subjects will be screened within 35 days before their dose of trial medication and reside at the Investigator site from the day before their dose (Day -1) until approximately 24 hours after dosing (Day 2). They will return for a follow-up visit on Day 8-9.

Part B will include up to 24 healthy subjects in up to 3 groups of 8 subjects (Groups B1-B3). Subjects will receive once-daily intranasal doses of Neumifil or placebo for 7 days. In each group, 6 subjects will receive Neumifil and 2 subjects will receive matching placebo.

The starting dose level (dose and dose regimen) for Group B1 will be decided after review of safety and tolerability data from at least 3 dose levels in Part A, and will be no higher than a dose that has previously been shown to cause no safety concerns in Part A . An additional dose level may be explored in 1 optional group of up to 8 subjects (Group B4).

Subjects will be screened within 35 days before their dose of trial medication and reside. at the Investigator site from the day before their first dose (Day -1) until about 24 hours after their last dose (Day 8). Subjects will attend an outpatient visit on Days 15-16. They will return for a follow-up visit on Days 21-23.

During the study, dose levels for study groups will be determined by a Safety Review Committee in accordance with criteria defined in the study protocol and the Investigator site operating procedures. Dose levels will only be increased if the safety and tolerability of previous dose levels are considered to be acceptable by the Safety Review Committee.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female volunteer, aged 18-60 years.
2. BMI (Quetelet index) in the range 18.0-30.9 kg/m2.
3. Able to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire trial.
4. Willingness to give written consent to participate after reading the information and consent form, and after having the opportunity to discuss the trial with the investigator or their delegate.
5. Agree to follow the contraception requirements of the trial
6. Agree not to donate blood or blood products during the study and for up to 3 months after the administration of the trial medication.
7. Spirometry readings (FEV1 and FVC) to be ≥ 80% of predicted value at the screening visit, calculated using National Health and Nutrition Examination Survey (NHANES) reference. If a subject's FEV1 or FVC is outside that range at the screening visit, the test may be repeated once on another day.
8. Registered with a General Practitioner (GP) in the UK (Part A only).
9. Willingness to give written consent to have data entered into The Overvolunteering Prevention System (TOPS).

Exclusion Criteria:

1. Woman who is pregnant or lactating, or pre-menopausal woman who is sexually active and not using a reliable method of contraception.
2. Clinically relevant abnormal medical history, physical findings, ECG, or laboratory values at the pre-trial screening assessment that in the opinion of the investigator could interfere with the objectives of the trial or the safety of the volunteer.
3. Presence or history of acute or chronic illness sufficient to invalidate the volunteer's participation in the trial or make it unnecessarily hazardous.
4. Presence or history of respiratory disease, including (but not limited to) asthma, chronic obstructive pulmonary disease (COPD), cystic fibrosis, emphysema, requiring acute or chronic medication.
5. Presence of nasal polyps or significant nasal abnormalities.
6. Symptoms of respiratory illness (including, but not limited to, runny nose, sore throat, sneezing, coughing or wheezing) at the screening visit or before dosing on Day 1.
7. Tympanic temperature > 37.5°C at the screening visit or before dosing on Day 1.
8. Impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease, or history of any psychotic mental illness.
9. History of psychiatric disease, as determine by the investigator.
10. History or presence of malignant disease.
11. Immune-suppressed status, resulting from either disease or medication, as determined by the investigator.
12. Presence or history of severe adverse reaction to any drug or the excipients of Neumifil.
13. Known allergy to tetracycline antibiotics.
14. Use of a prescription medicine (except HRT in female subjects), including oral contraceptives, during the 28 days before the first dose of trial medication, or use of an over-the-counter medicine, with the exception of acetaminophen (paracetamol) and vitamin or nutritional supplements, during the 7 days before the first dose of trial medication.
15. Receipt of an investigational product (including prescription medicines) as part of another clinical trial within the 3 months before admission to this study; in the follow-up period of another clinical trial at the time of screening for this study.
16. Receipt of a COVID-19 vaccine within 7 days before the first dose of trial medication, or anticipate receiving a COVID-19 vaccine within the 7 days after a (final) dose of trial medication.
17. Presence or history of drug or alcohol abuse, or regular intake of more than 14 units of alcohol weekly.
18. Use of cigarettes or nicotine-containing products during the 6 months before first dose of trial medication.
19. Blood pressure and heart rate in supine position at the screening examination outside the ranges: blood pressure 90-140 mm Hg systolic, 40-90 mm Hg diastolic; heart rate 40-100 beats/min. Triplicate measurements will be made (at least 2 min apart), and a mean value outside the above ranges will lead to exclusion. Repeat measurements (in triplicate) are permitted if values are borderline (ie values that are within 5 mm Hg for blood pressure or 5 beats/min for heart rate) or if requested by the investigator. Subjects can be included if the repeat value is within range or still borderline but deemed not clinically significant by the investigator.
20. QTcF value, of > 450 msec (men) or > 470 msec (women); or QRS duration

    ≥ 120 msec, measured on 12-lead ECG at the screening visit. Triplicate measurements will be made, and a mean value used to determine eligibility. A repeat (in triplicate) is also allowed on one occasion for determination of eligibility.
21. Possibility that the volunteer will not cooperate with the requirements of the protocol.
22. Positive test for hepatitis B surface antigen, hepatitis C or HIV. NOTE:

    participants with positive hepatitis C antibody owing to resolved disease can be included only if a hepatitis C ribonucleic acid (RNA) test is negative.
23. Positive test for SARS-CoV-2 (polymerase chain reaction; PCR) or suspected exposure to the SARS-CoV-19 virus during the 14 days before screening.
24. Loss of more than 400 mL blood during the 3 months before the trial, eg as a blood donor.
25. Objection by GP to volunteer entering trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Kitson, Study Director — gkitson@propharmapartners.uk.com
Locations (1):
- Hammersmith Medicines Research (HMR), London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a first in human study in healthy participants at a single site in the UK. The first participant was screened on 07 October 2021 and the last participant visit was on 05 April 2022.
Groups:
- Part A Placebo All Groups: Placebo single dose for all groups
- Part A1 Neumifil 0.028mg: Neumifil 0.028mg single dose
- Part A2 Neumifil 0.085mg: Neumifil 0.085mg single dose
- Part A3 Neumifil 0.28mg: Neumifil 0.28mg single dose
- Part A4 Neumifil 0.885mg: Neumifil 0.885mg single dose
- Part A5 Neumifil 2.8mg: Neumifil 2.8mg single dose
- Part B Placebo All Groups: Placebo once daily for 7 days for all.groups
- Part B1 Neumifil 0.28mg: Neumifil 0.28mg once daily for 7 days
- Part B2 Neumifil 0.885mg: Neumifil 0.885mg once daily for 7 days
- Part B3 Neumifil 2.8mg: Neumifil 2.8mg once daily for 7 days
Period: Overall Study
Arm/Group | Part A Placebo All Groups | Part A1 Neumifil 0.028mg | Part A2 Neumifil 0.085mg | Part A3 Neumifil 0.28mg | Part A4 Neumifil 0.885mg | Part A5 Neumifil 2.8mg | Part B Placebo All Groups | Part B1 Neumifil 0.28mg | Part B2 Neumifil 0.885mg | Part B3 Neumifil 2.8mg
Started | 12 | 4 | 4 | 4 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 12 | 4 | 4 | 4 | 6 | 6 | 5 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A Placebo All Groups: Placebo will be administered intranasally using an Aptar deliver system. Each dose will consist of 0.5ml to each nostril.
- Part A1 Neumifil 0.028mg; Part A3 Neumifil 0.28mg: Neumifil 0.028mg as a single dose administered intranasally using an Aptar delivery system. Each dose will consist of 0.5ml to each nostril.
- Part A2 Neumifil 0.085mg; Part A4 Neumifil 0.885mg: Neumifil 0.085mg as a single dose administered intranasally using an Aptar delivery system. Each dose will consist of 0.5ml to each nostril.
- Part A5 Neumifil 2.8mg: Neumifil 2.8 mg as a single dose administered intranasally using an Aptar delivery system. Each dose will consist of 0.5ml to each nostril.
- Part B Placebo All Groups: Placebo will be administered intranasally once daily for 7 days using an Aptar delivery system. Each dose will consist of 0.5ml to each nostril.
- Part B1 Neumifil 0.28mg: Neumifil 0.28mg will be administered intranasally once daily for 7 days using an Aptar delivery system. Each dose will consist of 0.5ml to each nostril.
- Part B2 Neumifil 0.885mg: Neumifil 0.885mg will be administered intranasally once daily for 7 days using an Aptar delivery system. Each dose will consist of 0.5ml to each nostril.
- Part B3 Neumifil 2.8mg: Neumifil 2.8mg will be administered intranasally once daily for 7 days using an Aptar delivery system. Each dose will consist of 0.5ml to each nostril.
- Total: Total of all reporting groups
Arm/Group | Part A Placebo All Groups | Part A1 Neumifil 0.028mg | Part A2 Neumifil 0.085mg | Part A3 Neumifil 0.28mg | Part A4 Neumifil 0.885mg | Part A5 Neumifil 2.8mg | Part B Placebo All Groups | Part B1 Neumifil 0.28mg | Part B2 Neumifil 0.885mg | Part B3 Neumifil 2.8mg | Total
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (12.16) | 34.0 (5.89) | 35.0 (14.85) | 31.5 (17.23) | 32.2 (12.94) | 27.7 (3.67) | 41.2 (15.32) | 38.8 (15.51) | 32.7 (12.19) | 38.3 (13.53) | 35.6 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 1 | 3 | 2 | 2 | 1 | 1 | 1 | 16
  Male | 9 | 3 | 3 | 3 | 3 | 4 | 4 | 5 | 5 | 5 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 12 | 4 | 4 | 4 | 6 | 6 | 6 | 5 | 5 | 6 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 12 | 4 | 4 | 4 | 6 | 6 | 6 | 6 | 6 | 6 | 60

OUTCOME MEASURES:

1. Primary Outcome: Part A Treatment Emergent Adverse Events
Description: Number of participants with Treatment Emergent Adverse Events
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Groups:
- Part A4 0.Neumifil 0.885mg: Neumifil 0.085mg as a single dose administered intranasally using an Aptar delivery system. Each dose will consist of 0.5ml to each nostril.
Arm/Group | Part A Placebo All Groups | Part A1 Neumifil 0.028mg | Part A2 Neumifil 0.085mg | Part A3 Neumifil 0.28mg | Part A4 0.Neumifil 0.885mg | Part A5 Neumifil 2.8mg
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 6 | 6
Participants | 4 | 3 | 2 | 3 | 5 | 5

2. Primary Outcome: Part B: Treatment Emergent Adverse Events
Description: Number of participants with Treatment Emergent Adverse Events
Time Frame: 14 days after last dose
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Placebo All Groups | Part B1 Neumifil 0.28mg | Part B2 Neumifil 0.885mg | Part B3 Neumifil 2.8mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 5 | 6 | 5 | 6

3. Primary Outcome: Part A: Clinically Significant Changes in Safety Tests
Description: Number of participants with clinically significant changes in:vital signs (heart rate, blood pressure, respiratory rate, pulse oximetry and temperature), 12-lead electrocardiogram (ECG), Forced expiratory volume in 1 second (FEV1), Forced vital capacity (FVC), physical examination, nasal examination, laboratory safety tests (haematology, biochemistry and urinalysis), tolerability questionnaire
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Part A Placebo All Groups | Part A1 Neumifil 0.028mg | Part A2 Neumifil 0.085mg | Part A3 Neumifil 0.28mg | Part A4 0.Neumifil 0.885mg | Part A5 Neumifil 2.8mg
Number analyzed (Participants) | 12 | 4 | 4 | 4 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part B:Clinically Significant Changes in Safety Tests
Description: Number of participants with clinically significant changes in: vital signs (heart rate, blood pressure, respiratory rate, pulse oximetry and temperature), 12-lead electrocardiogram (ECG), FEV1, FVC, physical examination, nasal examination, laboratory safety tests (haematology, biochemistry and urinalysis), tolerability questionnaire
Time Frame: 14 days after last dose
Measure: Count of Participants; unit: Participants
Arm/Group | Part B Placebo All Groups | Part B1 Neumifil 0.28mg | Part B2 Neumifil 0.885mg | Part B3 Neumifil 2.8mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 1 | 0 | 0 | 0

5. Other Pre Specified Outcome: SARS-CoV-2 Infection Test
Description: SARS-CoV-2 infection test
Time Frame: Screening, before first dose, Day 8 (Part B only), follow-up (Part A: Day 8 to 9); Part B: Day 21 to 23)
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Part B: Immunoglobulin A and G (IgA and IgG) Concentrations
Description: Part B: Immunoglobulin A and G (IgA and IgG) concentrations specific for Neumifil
Time Frame: Blood samples before first dose, follow-up (Day 21 to 23)
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Part A: Plasma Concentration of Neumifil
Description: Part A: Plasma concentration of Neumifil
Time Frame: Day 1 after single dose
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Part B:Plasma Concentration of Neumifil
Description: Part B:Plasma concentration of Neumifil
Time Frame: Day 1 after dosing, Day 7
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 7 days after single dose groups (all Part A groups) and 14 days after the last dose for multiple dose groups (all Part B groups)
Arm/Group | Part A Placebo All Groups | Part A1 Neumifil 0.028mg | Part A2 Neumifil 0.085mg | Part A3 Neumifil 0.28mg | Part A4 Neumifil 0.885mg | Part A5 Neumifil 2.8mg | Part B Placebo All Groups | Part B1 Neumifil 0.28mg | Part B2 Neumifil 0.885mg | Part B3 Neumifil 2.8mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/4 | 0/4 | 0/4 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/4 | 0/4 | 0/4 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/12 | 3/4 | 2/4 | 3/4 | 5/6 | 5/6 | 5/6 | 6/6 | 5/6 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Placebo All Groups (N=12) | Part A1 Neumifil 0.028mg (N=4) | Part A2 Neumifil 0.085mg (N=4) | Part A3 Neumifil 0.28mg (N=4) | Part A4 Neumifil 0.885mg (N=6) | Part A5 Neumifil 2.8mg (N=6) | Part B Placebo All Groups (N=6) | Part B1 Neumifil 0.28mg (N=6) | Part B2 Neumifil 0.885mg (N=6) | Part B3 Neumifil 2.8mg (N=6)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 2 (2) | 2 (4) | 4 (5) | 4 (9) | 3 (5) | 4 (4) | 3 (5) | 3 (6)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Product after taste (Product Issues) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 2 (2) | 4 (4) | 3 (3) | 2 (2)
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cather site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT05093530/Prot_SAP_000.pdf